CLINICAL TRIAL: NCT03532308
Title: Assessing the Clinical Response of Prostate Cancer to a Fermented Soy Extract
Brief Title: Nutrition and Prostate Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to meet recruitment goals.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000020868
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Results first posted 2021-05-06 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Prostate Cancer
Keywords: Fermented Soy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Daily Fermented Soy (two 12.5g packets/day) (~1 ounce/day) taken between the time of enrollment and radical prostatectomy (RP). Clinical assessment of both groups will take place 1) at baseline, and 2) just prior to RP, estimated at between 4 and 10 weeks from baseline/enrollment. Length of time in the study will vary for each subject, depending on how far out their prostatectomy will occur; all prostatectomies will be scheduled to occur between 4-10 weeks post-baseline.
  Interventions: Drug: Fermented Soy
- Placebo (Placebo Comparator): Daily (matched dose) taken between the time of enrollment and radical prostatectomy (RP). Clinical assessment of both groups will take place 1) at baseline, and 2) just prior to RP, estimated at between 4 and 10 weeks from baseline/enrollment. Length of time in the study will vary for each subject, depending on how far out their prostatectomy will occur; all prostatectomies will be scheduled to occur between 4-10 weeks post-baseline.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fermented Soy — Two 12.5g packets/day) (~1 ounce/day) taken between the time of enrollment and radical prostatectomy (RP). Time can be between 4 and 10 weeks.
  Other Names: Q-CAN Plus
  Arms: Intervention
Other: Placebo — A placebo compliment to the active intervention with identical packaging and labeling will be used.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of Fermented Soy vs. placebo in 72 adults with localized prostate cancer prior to radical prostatectomy.

DETAILED DESCRIPTION:
This is a parallel group, double-blind, randomized clinical trial with two arms. The primary aim is to assess the efficacy of Fermented Soy vs. placebo in 72 adults with prostate cancer. This study has 1 primary aim and 3 (1a thru 1c) sub aims. Aim 1 is to assess the effect of Fermented Soy (QC) on PSA (prostate specific antigen) In parallel, in Aims 1a-1c will assess tumor-specific effects of QC:

Aim 1a: Identifying the anti-tumor effects of QC. This will be done by culturing multiple human cancer cell lines with QC at a range of concentrations, followed by readouts at different time points, of tumor cell apoptosis, proliferation, and senescence.

Aim 1b: Identify a hierarchy of tumors that are responsive to QC. From the data in aim one an attempt will be made to identify a hierarchy of anti-tumor effects.

Aim 1c: Investigate the signaling pathways in tumor cells that are modified by QC. To do this, full genomic profiling will be conducted for breast and prostate tumor cell lines, and will be done in conjunction with analysis of the relevant signaling pathways, and will include P53 and P21 activation pathways.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified Prostate Cancer (at any stage)
* Scheduled to be treated by radical prostatectomy within the next 4-10 weeks
* Understanding and willingness to provide consent

Exclusion Criteria:

* Previous (within 6 months of enrollment) or concurrent hormonal therapy or chemotherapy; specifically, treatment with 5-alpha reductase inhibitors (finasteride and dutasteride)
* History of hormone dependent malignancies
* Concomitant thyroid disease or currently taking thyroid hormone replacement medication
* Current high-dose soy consumption, micronutrient, or herbal supplements, on soy or vegetarian nutrition, or any other extreme dietary habits
* Current or past history of any liver or pancreas disease
* History of allergy or hypersensitivity to soy-containing products
* Malabsorption conditions that might interfere with absorption of the investigational product

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2019-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Yale University, New Haven, Connecticut
  - Yale New Haven Health- Lawrence + Memorial Hospital, New London, Connecticut
  - South County Hospital, Wakefield, Rhode Island

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Placebo
Started | 10 | 9
Completed Assessments | 9 | 7
Completed | 10 | 8
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants enrolled and randomized to a treatment arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Placebo | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (6.9) | 62.9 (6.4) | 61.7 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19
CAPRA Score [Count of Participants; unit: Participants] — The CAPRA score is a measure of prostate cancer risk that ranges from 0 - 10. A CAPRA score of: 0 to 2 indicates low-risk, 3 to 5 indicates intermediate-risk, 6 to 10 indicates high-risk. For the purposes of this study, the low-risk and intermediate-risk groups were combined as part of the randomization stratification.
  Participants
    0-5: Low/Intermediate risk | 5 | 5 | 10
    6-10: High risk | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Prostate-specific Antigen (PSA)
Description: The PSA test measures the level of PSA in a man's blood. For this test, a blood sample is sent to a laboratory for analysis. The results are usually reported as nanograms of PSA per milliliter (ng/mL) of blood. The PSA range of scores and interpretation are as follows: Normal PSA Levels: 0 - 4 ng/mL, Slightly Elevated PSA: 4 - 10 ng/mL, Moderately Elevated PSA: 10 - 20 ng/mL, Highly Elevated PSA: 20+ ng/mL. Interpretation of these scores is also based on the age of the inidividual.
Time Frame: Greater than or equal to 4 weeks (up to 10 weeks)
Population: Intention to treat analysis population.
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 10 | 9
ng/mL
  Baseline | 8.97 (1.10) | 8.66 (1.16)
  Up to 10 Weeks | 8.11 (1.12) | 8.92 (1.21)
Statistical Analysis 1: Comparison: Intervention vs Placebo; Test type: Superiority; p = 0.76, Mixed Models Analysis — This is for the effect of treatment with time, risk stratification and treatment*time interaction in the model

2. Secondary Outcome: Gleason Score
Description: Pathological investigation of the removed prostate gland will include the assessment of biopsy-proven, index prostate cancer lesion will lead to the analysis of any modulation of PCa grade (Gleason score) compared to preoperative biopsies. The Gleason Score is interpreted as follows: 3+4 (Prognosis = Good), 4+3 (Prognosis = Likely to Spread), 8 - 10 (Prognosis = Likely to Spread Rapidly).
Time Frame: Greater than or equal to 4 weeks (up to 10 weeks)
Population: Participants that were available for assessment at the end of treatment/study.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 8 | 8
Participants
  3+4 (Prognosis = Good) | 7 | 5
  4+3 (Prognosis = Likely to Spread) | 0 | 2
  8 - 10 (Prognosis = Likely to Spread Rapidly) | 1 | 1

3. Secondary Outcome: PCa Tissue Telomeric DNA Length
Description: Analysis of telomere length in research samples of human peripheral blood mononuclear cells reveals that telomere length decreases with increased replication of cells, reflecting the replicative history of those cells.
Time Frame: Greater than or equal to 4 weeks (up to 10 weeks)
Population: These data were not collected due to early termination of the study.
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Cancer of the Prostate Risk Assessment (CAPRA-S) Score Change
Description: Post surgical/post intervention CAPRA score will be used for comparison with baseline (screening) value. The CAPRA score can range from 0 to 10 where: a score of 0 to 2 indicates low-risk, 3 to 5 indicates intermediate-risk, and 6 to 10 indicates high-risk.
Time Frame: Baseline to final visit (up to 10 weeks)
Population: Per protocol change in scores from baseline in those with complete data at baseline and end of study/treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 8 | 8
units on a scale | -1.3 (0.9) | -1.4 (1.3)

5. Secondary Outcome: Cell Cycle Progression Score
Description: Assessment of prostate cancer mRNA can be determined from PCa tissue. Cell cycle progression score assessment of PCa mRNA is a novel RNA expression-based assay that directly measures tumor cell growth characteristics in order to stratify patients with localized PCa according to disease aggressiveness.
Time Frame: Greater than or equal to 4 weeks (up to 10 weeks)
Population: These data were not collected due to early termination of the study.
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Functional Assessment of Cancer Therapy - Prostate (FACT-P v4©)
Description: Quality of life assessment for men with PCa will be assessed with the Functional Assessment of Cancer Therapy - Prostate (FACT-P v4©). The FACT-P contains 39 items that use a 0-4 rating scale. The highest possible score is 156 (lowest possible score = 0). The total score is an indication of overall quality of life where the higher scores indicate better quality of life.
Time Frame: Greater than or equal to 4 weeks (up to 10 weeks)
Population: Presented are data for all participants with complete data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 10 | 9
units on a scale
  Baseline | 121.50 [104.47 to 138.53] | 128.44 [118.07 to 138.82]
  End of Study (up to 10 weeks): number analyzed (Participants) | 10 | 8
  End of Study (up to 10 weeks) | 126.00 [113.04 to 138.96] | 123.25 [112.79 to 133.71]

ADVERSE EVENTS:
Time Frame: Up to 10 weeks
Arm/Group | Intervention | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/9
Other Adverse Events (participants affected / at risk) | 3/10 | 1/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=10) | Placebo (N=9)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Unrelated hospitalization where participant experienced an Aortic Aneurysm and presented with Pneumonia.
Aortic Aneurysm (Cardiac disorders) | 1 (1) | 0 (0) — Unrelated hospitalization where participant experienced an Aortic Aneurysm and presented with Pneumonia.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=10) | Placebo (N=9)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nausea/Dizzyness (Nervous system disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/08/NCT03532308/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT03532308/SAP_001.pdf